CLINICAL TRIAL: NCT06782776
Title: Retrospective and Prospective Study on the Role of Doppler Echoflowmetry in Defining Risk Factors for the Development of Complications in Twin Pregnancies
Brief Title: Role of Doppler Echoflowmetry to Define Risk Factors for the Development of Complications in Twin Pregnancies
Acronym: TWINS
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: TWINS
Record Dates: First submitted 2024-12-03; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-10

CONDITIONS: Twin Pregnancy, Antepartum Condition or Complication
Keywords: Doppler echflowmetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to evaluate the outcomes of twin pregnancies referred to our center, in order to understand whether the use of different guidelines over time, with more systematic follow-up timing, has improved their management by reducing adverse events. All this would provide us with useful information for a better understanding of the effects of twinhood on pregnancy outcomes, so that we have more accurate information in counseling with patients.

DETAILED DESCRIPTION:
The study is retrospective and prospective. Patients for whom twin pregnancy was monitored at the outpatient clinics of the division of Obstetrics and Prenatal Age Medicine, a regional referral center for the management of complicated pregnancies, will be enrolled.

Only those patients for whom the delivery was carried out at the same facility will be considered. This first phase will be necessary to obtain specific information about the complication rate and course of twin pregnancies that over the past 15 years (2005 to present) have been afferent at our facility. All patients will undergo the ultrasound evaluations required by the normal care protocols for twin pregnancies (biweekly checks if monochorionic or monthly if bicorionic) until 2026.

In addition to the standard ultrasound monitoring, an instrumental assessment will then be performed by means of the USCOM 1A ® technique, an ultrasound instrument that, by inputting the patient's height and weight, is able to calculate, thanks to internal algorithms, the diameter of the aortic valve and the blood flow through the valve itself. In addition, the peak pulsatility of the maternal ophthalmic artery will be assessed by Doppler ultrasound technique, which appears to be predictive of the risk of developing preeclampsia. In addition to the normal ultrasound evaluation provided by the current care procedure, an echocardiographic acquisition of the fetal heart by STRAIN technique will be performed.

Two-dimensional strain is based on the acquisition of a typical myocardial pattern (called finger print), which can be followed during the cardiac cycle. In other words, the software recognizes a small piece of tissue, evaluating its strain. Because of its angle-independence, two-dimensional strain allows global and segmental assessment of myocardial contractility, both longitudinal and radial. In these patients, strain would have the ability to detect a contractility deficit evidenced by a reduction in peak systolic strain and strain rate, which, as already demonstrated in adults, distinguishes areas of increased fibrosis, myocyte loss, and myocardial fiber reorganization. Strain may also be useful in prognostic stratification of heart failure, distinguishing fetuses with particularly impaired contractile capacity.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Twin Pregnancy
* Ultrasound monitoring and delivery occurred at Policlinico S Orsola in Bologna, Italy
* Written informed consent form obtained from the patient

Exclusion Criteria:

* Completion of delivery at another facility
* Desire to undertake the Voluntary Interruption of Pregnancy
* Refusal to undergo instrumental monitoring and subsequent follow-up at our center

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will consist of patients with twin pregnancies, regardless of chorionicity, who access the Pregnancy at Risk outpatient clinic at our center to perform the specific diagnostic care pathway.
Sampling Method: Non-Probability Sample
Enrollment: 6600 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Consequences of twinning on maternal and fetal hemodynamics | up to 100 weeks
  Evaluation of the effects and consequences of twinning on maternal and fetal hemodynamics during pregnancy.

SECONDARY OUTCOMES:
Potential risk factors for the development of adverse maternal or fetal outcomes | up to 100 weeks
  Assessment of the presence of specific and potential risk factors for the development of adverse maternal or fetal outcomes
Assessment of the presence of any different outcomes in relation to the guidelines applied in the past | up to 100 weeks
  Compare the guidelines applied in the past with the results obtained from the outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Gianluigi Pilu, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy